CLINICAL TRIAL: NCT01514942
Title: Myo-inositol Versus D-chiro-inositol in the Treatment of Polycystic Ovary Syndrome and Insulin Resistance: Evaluation of Clinical, Metabolic, Endocrine and Ultrasound Parameters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: MIvsDCI_PCOS/IR
Record Dates: First submitted 2012-01-13; First posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: PCOS
Keywords: PCOS; Insulin resistance; Myo-inositol; D-chiro-inositol
MeSH Terms: conditions — Insulin Resistance | interventions — Inositol; Folic Acid; Manganese; Vitamin B 12

ARMS (2):
- Insulin resistant patients (Other)
  Interventions: Dietary Supplement: Myo-inositol + Folic acid; Dietary Supplement: D-chiro-inositol, manganese, folic acid, vit B12; Drug: Folic acid, vit B12
- Non-insulin resistant patients (Other)
  Interventions: Dietary Supplement: Myo-inositol + Folic acid; Dietary Supplement: D-chiro-inositol, manganese, folic acid, vit B12; Drug: Folic acid, vit B12

INTERVENTIONS:
Dietary Supplement: Myo-inositol + Folic acid — Myo-inositol (2g) Folic acid (200mcg) (2 per day)
  Arms: Insulin resistant patients
Dietary Supplement: Myo-inositol + Folic acid — Myo-inositol (2g) Folic acid (200mcg) (2 per day)
  Arms: Non-insulin resistant patients
Dietary Supplement: D-chiro-inositol, manganese, folic acid, vit B12 — D-Chiro-inositol (500 mg), manganese (1 mg), folic acid (200 mcg), vit B12 (1.25 mcg) (2 per day)
  Arms: Insulin resistant patients
Dietary Supplement: D-chiro-inositol, manganese, folic acid, vit B12 — D-chiro-inositol (500 mg), manganese (1 mg), folic acid (200 mcg), vit B12 (1.25 mcg) (2 per day)
  Arms: Non-insulin resistant patients
Drug: Folic acid, vit B12 — Folic acid (200 mcg), vit B12 (1.25 mcg) (2 per day)
  Arms: Insulin resistant patients
Drug: Folic acid, vit B12 — Folic acid (200 mcg), vit B12 (1.25 mcg) (2 per day)
  Arms: Non-insulin resistant patients

SUMMARY:
Insulin resistance has important implications in the pathogenesis of the polycystic ovary syndrome (PCOS) and insulin-sensitizing drugs are considered a useful therapeutic approach.

Reduction of insulin levels with administration of insulin sensitizing agents has been found to be beneficial in lowering both hyperinsulinemia, hyperandrogenemia, and restoring ovulation. Metformin alone or in combination with oral contraceptives (OCs) has been widely used in the long term treatment of women with PCOS in whom it modifies the ovarian morphology, improves intraovarian androgen levels, and enhances systemic and local insulin resistance. Despite to these beneficial effects, several side effects have been reported due to the long term administration of this drug.

In the recent years, inositol has found more and more space in the reproductive clinical practice. Indeed, inositol have been classified as "insulin sensitizing agent" and it is mainly used as a chronic treatment for PCOS. Inositol exists in 9 different isomers and in particular several studies on Myo-inositol and D-chiro-inositol were reported.

In this study myo-inositol versus D-chiro-inositol treatments were compared to placebo in women with PCOS and with or without insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Women fulfilled two out of three diagnostic criteria for PCOS

Exclusion Criteria:

* Women with pre-existing secondary endocrine disorders
* Women with personal history of hypertension, diabetes mellitus or cardiovascular disorders
* Women who received treatment with other drugs for the previous 6 months before entering the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Body Mass Index (BMI)
Menstrual cycle
Score acne (acne grading system by Cremoncini et al)
Score hirsutism (Ferriman-Gallwey score)
Alopecia
Oral Glucose Tolerance Test (OGTT)
Glucagon levels
C-peptide test
Myo-inositol serum concentration
D-chiro-inositol serum concentration
Luteinizing Hormone (LH), Follicle Stimulating Hormone (FSH), and Estradiol (E2) levels test
Prolactin (PRL) levels test
Thyroid-stimulating hormone (TSH), free thyroid hormone (fT3 and fT4), and alpha-1 antitrypsin (AAT) test
Total and free testosterone levels
Sex hormone binding globulin (SHBG) test
17-Hydroxyprogesterone (17-OHP) levels
Dehydroepiandrosterone (DHEA) and DHEA-sulfate (DHEAS) levels
delta 4-androstenedione levels
progesterone levels
Adrenocorticotropic Hormone (ACTH) stimulation test
Ovarian size and morphology
  Ovarian ultrasound scan for the assessment of size and morphology
Antral follicle counts
Stromal/Cortical ratio in the ovary
Endometrial thickness
  Transvaginal ultrasound measurement of endometrial thickness performed between day 3 and 5 of the menstrual cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto di Patologia Ostetrica e Ginecologica, Catania, Italy

REFERENCES:
- [Background] Costantino D, Minozzi G, Minozzi E, Guaraldi C. Metabolic and hormonal effects of myo-inositol in women with polycystic ovary syndrome: a double-blind trial. Eur Rev Med Pharmacol Sci. 2009 Mar-Apr;13(2):105-10. PMID 19499845
- [Background] Raffone E, Rizzo P, Benedetto V. Insulin sensitiser agents alone and in co-treatment with r-FSH for ovulation induction in PCOS women. Gynecol Endocrinol. 2010 Apr;26(4):275-80. doi: 10.3109/09513590903366996. PMID 20222840
- [Background] Larner J. D-chiro-inositol--its functional role in insulin action and its deficit in insulin resistance. Int J Exp Diabetes Res. 2002;3(1):47-60. doi: 10.1080/15604280212528. PMID 11900279
- [Background] Larner J, Brautigan DL, Thorner MO. D-chiro-inositol glycans in insulin signaling and insulin resistance. Mol Med. 2010 Nov-Dec;16(11-12):543-52. doi: 10.2119/molmed.2010.00107. Epub 2010 Aug 27. PMID 20811656